CLINICAL TRIAL: NCT03824288
Title: A Randomized Multicenter Trial of Ultrasound-Guided Aspiration of Peritonsillar Abscess Versus Conventional Landmark Technique
Brief Title: Ultrasound-Guided Aspiration of PTA vs Conventional Landmark Technique - a RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tobias Todsen (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Tobias Todsen, MD, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: VD-2018-361
Record Dates: First submitted 2019-01-23; First posted 2019-01-31 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Peritonsillar Abscess
MeSH Terms: conditions — Peritonsillar Abscess

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The landmark technique (Active Comparator): PTA a needle aspiration attempted according to the landmark technique is conducted. If the initial aspiration is unsuccessful, two additional attempts are made in the middle and lower pole of the tonsil.
  Interventions: Procedure: The landmark technique
- Ultrasound-guided aspiration (Experimental): An intraoral ultrasound is conducted with a Burr-Hole N11C5s transducer (BK Ultrasound) and if an abscess cavity is suspected, an ultrasound-guided aspiration is performed with an in-plane needle guide attached to guide the needle.
  Interventions: Diagnostic Test: Intraoral ultrasound

INTERVENTIONS:
Diagnostic Test: Intraoral ultrasound — The ultrasound transducer (either Hockey Stick or Burr-Hole N11C5s transducer from BK Ultrasound) is placed on the palatoglossal arch on the affected side and sweeped from the cranial to caudal end of the tonsil to look for an abscess cavity identified as a hypoechoic area with ill-defined margins.
  Arms: Ultrasound-guided aspiration
Procedure: The landmark technique — A 14G needle aspiration is inserted blindly in the superior tonsil pol where pus aspiration is attempted.
  Arms: The landmark technique

SUMMARY:
The study is a prospective randomized controlled trial conducted at two different centers at the Department of ORL - Head & Neck Surgery, Odense University Hospital and the Department of Otorhinolaryngology, Head and Neck Surgery & Audiology, Rigshospitalet.

The research question is:

In a group of patients referred to an otolaryngology department with objective findings of peritonsillar abscess, what are the effects of using intraoral ultrasound to diagnose and guide needle aspiration compared to the traditional landmark-based technique, when measured by the number of performed needle aspirations, procedure-related pain and days on sick leave?

The secondary outcomes measured are

* Number of hospitalization days
* Number of Quincy tonsillectomies
* Number of visits to an outpatient clinic
* Patient-reported outcome (measured using an 11-point numeric rating scale)

ELIGIBILITY:
Inclusion criteria:

* Patients referred to the Department of Otorhinolaryngology suspected for peritonsillar abscess
* Clinical findings of peritonsillar abscess by one of the following:

  1. Trismus
  2. Unilateral tonsillar/peritonsillar swelling

Exclusion criteria:

* Compromised airways or suspected retro / parapharyngeal abscess
* Needle aspiration of pus already performed (or participated in the study once earlier)
* Cannot understand the written information

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
needle aspirations | From date of randomization until the date of full recovery from the treated peritonsilar infection, assessed up to 1 months.
  total number of needle aspirations performed
proportion of succesfull needle aspirations | From date of randomization until the date of full recovery from the treated peritonsilar infection, assessed up to 1 months.
  proportion of needle aspirations with aspiration of pus
days on sick leave | From date of randomization until the date of full recovery from the treated peritonsilar infection, assessed up to 1 months.
  Total number of days on sick leave after first intervention

SECONDARY OUTCOMES:
Number of hospitalization days | From date of randomization until the date of full recovery from the treated peritonsilar infection, assessed up to 1 months.
Number of quincy tonsillectomies | From date of randomization until the date of full recovery from the treated peritonsilar infection, assessed up to 1 months.
Number of visits in outpatient clinic | Until full recovery from peritonsilar infection
Patient-reported outcome | From date of randomization until the date of full recovery from the treated peritonsilar infection, assessed up to 1 months.
  Patients are asked to choose one number, on a scale from 0 (no pain) to 10 (severe pain), corresponding to the intensity of their pain - meassured using a 11-point numeric rating scale (NRS-11).

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen, Copenhagen East
  - Odense University Hospital, Odense, Odense C

REFERENCES:
- [Derived] Todsen T, Stage MG, Michaelsen SH, Tolsgaard MG, Melchiors J, Madsen AR, Hahn CH, Godballe C. Protocol for a randomised clinical trial of transoral ultrasound versus standard of care in the diagnosis of peritonsillar abscess. Dan Med J. 2019 Nov;66(11):A5573. PMID 31686648